CLINICAL TRIAL: NCT01127594
Title: A Multi-Center Phase I Dose Escalation Trial to Evaluate Safety and Tolerability of Intra-Arterial Temozolomide for Patients With Advanced Extremity Melanoma Using Normothermic Isolated Limb Infusion
Brief Title: Evaluate Safety/Tolerability Intra-Arterial Temozolomide in Patients w/Extremity Melanoma by Isolated Limb Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Douglas Tyler (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Duke University (Other); M.D. Anderson Cancer Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Douglas Tyler, Professor of Surgical Oncology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020406
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Temozolomide — Dose level selection will proceed according to the modified Accelerated Titration Design. The starting dose will be TMZ 200mg/m2 x 0.09 BSA for the upper extremity and 200mg/m2 x 0.18 BSA for the lower extremity. We will enroll one-patient cohorts with dose doubling between cohorts until 1st occurrence of a ≥ CTC (Common Terminology Criteria) grade 2 adverse event. At that time, the present cohort and all future cohorts will be extended to enroll 3 to 6 patients.
  Other Names: Temodar

SUMMARY:
The purpose of this study is to determine the safety profile of intra-arterial temozolomide administration during Isolated Limb Infusion (ILI) by defining the dose limiting toxicities associated with this treatment. This study also aims to determine the maximum tolerated dose of intra-arterial administration of temozolomide during ILI that will be used in a phase II trial.

DETAILED DESCRIPTION:
1. The primary objective of this study is to determine the safety profile of intra-arterial temozolomide administration during Isolated Limb Infusion (ILI) by defining the dose limiting toxicities associated with this treatment and to determine the maximum tolerated dose of intra-arterial administration of temozolomide during ILI that will be used in a phase II efficacy trial.
2. Population will include patients who have undergone a previous Melphalan based regional therapy for which they did not respond optimally and present with persistent, progressive, or recurrent disease. Study activities include tumor tissue sampling, blood sampling, and subjects will undergo an Isolated Limb Infusion.
3. To define both response in-field (area of the limb below the tourniquet) and out-of-field (any area outside the tourniquet) in patients treated with temozolomide based ILI. Response in this trial will be defined by the RECIST criteria (CR, PR, SD, PD at 12 weeks post ILI). A CR rate of 20% would be considered as preliminary evidence of a promising approach in this group of patients that have had a previous melphalan regional treatment. ILI with melphalan has a complete response rate of approximately 35% in naïve patients and 20% in patients who have previously received melphalan based regional therapy.

To assess if the proposed treatment has any effect on quality of life as measured by the Functional Assessment of Cancer Therapy - Melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have undergone a previous Melphalan based regional therapy for which they did not respond optimally and present with persistent, progressive, or recurrent disease.
2. Patient must be 18 years of age or older.
3. Patient must have an ECOG status of 0-1.
4. Patient must have histologically proven primary or recurrent extremity melanoma, stage IIIB, IIIC, or IV
5. Patients with Stage IIIC disease must either have had regional lymph nodes previously removed or will have them removed at the time of regional treatment.
6. Patients with Stage IV disease must have had all distant disease resected at least 30 days prior to regional treatment.
7. Disease to be treated by ILI must be distal to the planned site of tourniquet placement
8. Patient's disease must be bi-dimensionally measurable by caliper or radiological method as defined in the RECIST criteria.
9. Patient must have adequate bone marrow, liver and renal function
10. Patient must have a palpable femoral/radial pulse in the affected extremity.
11. Recovery from relevant toxicity prior to first study drug administration.
12. Patients must have a life expectancy of > 6 months.
13. Ability to read and understand English and the ability to complete paper +/- electronic survey assessments.

Exclusion Criteria:

1. Cardiac disease: Congestive heart failure > class II NYHA.
2. Known brain metastasis.
3. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
4. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
5. Active clinically serious infection > CTCAE Grade 2.
6. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
7. Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of administration of TMZ
8. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of administration of TMZ.
9. Serious non-healing wound, ulcer, or bone fracture.
10. Major surgery or significant traumatic injury within 30 days of ILI.
11. Evidence or history of bleeding diathesis or coagulopathy.
12. Antineoplastic therapy, radiotherapy, or any other investigational drug within 30 days prior to first study drug administration.
13. Patients with symptoms or signs of vascular insufficiency. Specifically, patients with any history of blood clots or lifestyle altering ischemic peripheral vascular disease will be excluded.
14. History of allergic reactions and/or hypersensitivity to TMZ.
15. Psychiatric conditions or diminished capacity that could compromise the giving of informed consent, or interfere with study compliance.
16. Pregnant or nursing women are not eligible for this study. Patients of reproductive potential must agree to use an effective method of birth control when undergoing treatments with known or possible mutagenic or teratogenic effects. All female participants of child-bearing potential must have a negative serum pregnancy test within two weeks of patient registration. Please note: use of contraception, including surgical procedures such as vasectomy or tubal ligation DO NOT eliminate the need for administering pregnancy testing.
17. Current treatment, or treatment in the previous 24 months, for another non-melanoma malignancy.
18. Unable to return at the regular required intervals for reassessment, or study drug administration.
19. Patients with known heparin induced thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety Profile of intra-arterial temozolomide and maximum tolerated dose of temozolomide | 12 Weeks
  To determine the safety profile of intra-arterial temozolomide administration during Isolated Limb Infusion (ILI) by defining the dose limiting (DLT) and non dose limiting toxicities associated with this treatment.
  To determine the maximum tolerated dose (MTD) for intra-arterial administration of temozolomide during ILI that will be used in a phase II efficacy trial.

SECONDARY OUTCOMES:
To define tumor response in field in patients treated with temozolomide | Until disease progression or death
  To define both response in-field (area of the limb below the tourniquet) and out-of-field (any area outside the tourniquet) in patients treated with temozolomide based ILI at the MTD dose. Response in this trial will be defined by the RECIST criteria (CR, PR, SD, PD at 12 weeks post ILI). A CR rate of 20% would be considered as preliminary evidence of a promising approach in this group of patients that have had a previous melphalan regional treatment. To assess if the proposed treatment has any effect on quality of life as measured by the Functional Assessment of Cancer Therapy - Melanoma.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Tyler, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas